CLINICAL TRIAL: NCT03784703
Title: Efficacy of Atorvastatin Versus Rosuvastatin on LV Function and Inflammatory Biomarkers in Type 2 Diabetic Patients With Dyslipidemia
Brief Title: Type 2 Diabetic Patients Maintained on Statin Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Damanhour University (Other)
Collaborators: Tanta University (Other)
Responsible Party: Principal Investigator, Rehab Werida, Clinical Pharmacy Lecturer, Damanhour University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Statin Therapy
Record Dates: First submitted 2018-12-13; First posted 2018-12-24 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Dyslipidemia Associated With Type II Diabetes Mellitus
Keywords: Adiponectin; Sortilin; Leptin; Dyslipidemia; Diabetes type II; Rosuvastatin; Atorvastatin
MeSH Terms: conditions — Dyslipidemias; Diabetes Mellitus, Type 2 | interventions — Atorvastatin; Tablets; Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: 160 patients were randomly assigned to receive either 40 mg per day atorvastatin tablets (ATROVA group, n= 80) or 10 mg per day Rosuvastatin tablets (ROSUVA group, n= 80) as recommended in NCEP ATP III (21). Patients included in the study were maintained on oral hypoglycemic agents (OHA) according to their treatment regimen.
Who Masked: Participant, Investigator
Masking Description: prospective, double blind trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atrovastatin (Experimental): atorvastatin (40 mg per day) for 6 months
  Interventions: Drug: Atorvastatin 40 Mg Oral Tablet
- Rosuvastatin (Experimental): Rosuvastatin (10 mg per day) for 6 months
  Interventions: Drug: Rosuvastatin 10 Mg Oral Tablet

INTERVENTIONS:
Drug: Atorvastatin 40 Mg Oral Tablet — 40 mg per day atorvastatin (ATROVA group, n= 80) for 6 months
  Other Names: Atorvastatin 40mg tablet per day
  Arms: Atrovastatin
Drug: Rosuvastatin 10 Mg Oral Tablet — 10 mg per day rosuvastatin (ROSUVA group, n= 80) for 6 months
  Other Names: Resovastatin 10 mg daily
  Arms: Rosuvastatin

SUMMARY:
Patients with diabetes mellitus (DM) are at increased risk of atherosclerotic cardiovascular disease (ACVD). The achievement of the LDL-C target with statins for the reduction of ACVD risk is recommended. However, the risk is still present. Therefore, we investigated the impact of high sensitivity C-reactive protein (hsCRP), sortilin, adiponectin and leptin biomarkers that linking inflammatory hypothesis of diabetes mellitus and atherosclerosis in diabetic patients treated with rosuvastatin and atrovastatin. Methods: Based on exclusion criteria, 150 type 2 diabetic patients were eligible and randomly assigned to receive either 40 mg per day atorvastatin (ATROVA group, n= 80) or 10 mg per day rosuvastatin (ROSUVA group, n= 80) for 6 months.

DETAILED DESCRIPTION:
a prospective, double blind trial, conducted between January 2018 and January 2020. Participants were enrolled if they had moderate cardiovascular risk (Framingham risk score of 10-20%), in other words 2 or more major risk factors for coronary artery disease (CAD), and LDL-cholesterol level ≥100 mg/dl. All patients gave informed consent before entering the study. Of 150 patients were randomly assigned to receive either 40 mg per day atorvastatin tablets (ATROVA group, n= 80) or 10 mg per day Rosuvastatin (Rosuvastatin Calcium®, Chemipharm Co. Cairo, Egypt) tablets (ROSUVA group, n= 80) as recommended in NCEP ATP III (21). Patients included in the study were maintained on oral hypoglycemic agents (OHA) according to their treatment regimen. Clinical and biochemical assessment was done at baseline and after 6 months. Serum High-sensitivity CRP (hsCRP), sortilin, Adiponectin and Leptin level was determined using ELISA Kit. Blood pressure (BP) and anthropometrical parameters, such as body-mass index (BMI) were calculated using the equation (BMI = weight (kg)/height (m2). Blood pressure was measured twice, after keeping participants in a sitting position for 15 min. The mean value of two consecutive measurements with 5 min intervals was used for study purposes. HbA1c% was determined by ion exchange method. Serum triglycerides (TGs), total cholesterol (TCH), and high-density lipoprotein cholesterol (HDL-C) were determined colorimetrically. Low-density lipoprotein-cholesterol (LDL-C) was calculated according to Friedewald formula. Atherogenic Index (AI) is calculated through the following: Atherogenic Index = TCH/HDL-C as TCH/HDL-C ratio is an excellent CVD risk predictor and a good biomarker for deciding on the intensity and the need for therapeutic intervention.

ELIGIBILITY:
Inclusion Criteria:

* type II diabetic patients with hypercholesterolemia

Exclusion Criteria:

* liver impairment,
* renal insufficiency,
* coronary artery disease,
* metabolic disorders,
* type I diabetes,
* autoimmune diseases, cancer, infection,
* use of anti-inflammatory drugs,
* recent major surgery,
* weight-loss or modified anti-hypertensive medications 12 weeks or less prior to enrolment,
* ongoing or previous use of lipid-lowering medications (including other statins, fibric acid derivatives, nicotinic acid, cholestyramine, ezetimibe or omega-3 fatty acids) and contraindications to the use of statins.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
hs-CRP (pg/mL) | 6 months
  biomarkers that linking the inflammatory hypothesis with diabetes mellitus and atherosclerosis.
sortilin (ng/mL) | 6 months
  Serum Level
adiponectin (ng/mL) | 6 months
  Serum Level
leptin (ng/mL) | 6 months
  Serum Level

SECONDARY OUTCOMES:
glucose level | 6 months
  fasting blood glucose (FBG) (mg/mL)
glycated hemoglobin | 6 months
  glycated hemoglobin (Hb A1c%)
total cholesterol | 6 months
  TCH: total cholesterol (mg/dL)
low density lipoprotein-cholesterol | 6 months
  LDL-C: low density lipoprotein-cholesterol (mg/dL), HDL-C: high density lipoprotein-cholesterol (mg/dL); Triglycerides (mg/dL).
high density lipoprotein-cholesterol | 6 months
  HDL-C: high density lipoprotein-cholesterol (mg/dL); Triglycerides (mg/dL).
Triglycerides | 6 months
  Triglycerides (mg/dL).

CONTACTS AND LOCATIONS:
Overall Officials: Rehab Werida, Lecturer, Study Director — Damanhour University
Locations (1):
- Tanta University Hospital, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krysiak R, Zmuda W, Okopien B. The effect of simvastatin-ezetimibe combination therapy on adipose tissue hormones and systemic inflammation in patients with isolated hypercholesterolemia. Cardiovasc Ther. 2014 Apr;32(2):40-6. doi: 10.1111/1755-5922.12057. PMID 24354929